CLINICAL TRIAL: NCT01777490
Title: Helping Invested Families Improve Veterans Experiences Study (HI-FIVES)
Brief Title: Helping Invested Families Improve Veterans Experiences Study
Acronym: HI-FIVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 11-345
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Caregiver; Disabled Veterans; Referred to Long-term Care; Residing at Home; Hospice Ineligible
Keywords: Caregivers - Not professionals; Frail Elderly; Long-term Care; Quality of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistant conducting follow-up interviews is blinded as to dyad arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Control - Caregiver (Active Comparator): Caregivers in the control arm will be referred to the VA Caregiver Support Program (usual care), as a resource for them as they care for the patient in the home.
  Interventions: Behavioral: Helping Invested Families Improve Veterans Experiences - Control
- Arm 2: HI FIVES - Caregiver (Experimental): Caregivers will take part in three phone training sessions and will attend four group training sessions at the VA. They will also be given the option of participating in 2 booster phone training sessions post-group sessions. Caregivers will be asked to provide one in-person (baseline) and three phone assessments (3, 9, and 15 months). Patients will also be enrolled and contact will be limited to assessments
  Interventions: Behavioral: Helping Invested Families Improve Veterans Experiences - HI FIVES
- Arm 1: Control - Patient (Active Comparator): The patient of each caregiver will also be enrolled and contact will be limited to assessments.
  Interventions: Behavioral: Helping Invested Families Improve Veterans Experiences - Control
- Arm 2: HI-FIVES - Patient (Experimental): The patient of each caregiver will also be enrolled and contact will be limited to assessments.
  Interventions: Behavioral: Helping Invested Families Improve Veterans Experiences - HI FIVES

INTERVENTIONS:
Behavioral: Helping Invested Families Improve Veterans Experiences - Control — Usual care will be the Veteran patient care and caregiver support that are normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This process entails the patient and caregiver work with the social worker assigned to the patient to obtain home and community based care (HCBC) services. The patients in the usual care group will be free to seek medical, psychological, social support, and social services that are available through VAMCs or any other source. In addition to this, caregivers in the usual care arm will be told about the caregiver support programs in the VHA and the caregiver will receive the national VA caregiver hotline phone number. The information provided mirrors efforts to support caregivers in the VA nationally and new standards of care for VA caregivers. This will be the only contact with the usual care subjects besides the scheduled data collection assessments.
  Other Names: Control
  Arms: Arm 1: Control - Caregiver; Arm 1: Control - Patient
Behavioral: Helping Invested Families Improve Veterans Experiences - HI FIVES — In addition to the usual care activities outline in the Control arm, Caregivers in the HI-FIVES group will receive three individual calls with a nurse educator to address topics he/she identified as being the highest priority learning areas. The calls will be tailored to the individual needs of Veteran-caregiver dyad. After the phone calls, caregivers will participate in four evidence-based group sessions aimed to improve clinical care skills, psychological care skills, and support-seeking skills. The curriculum will be delivered by a trained nurse educator and the PI and VA Caregiver Support Staff. The sessions will be targeted to address common needs of Veterans and their caregivers. After the final group session, there will be two optional booster calls at one and three months. Four assessments in all will be collected, baseline (in person), and at 3, 9, and 15 months (by phone).
  Other Names: Experimental
  Arms: Arm 2: HI FIVES - Caregiver; Arm 2: HI-FIVES - Patient

SUMMARY:
The purpose of this study is to evaluate a caregiver skill training program (HI-FIVES), offered as a part of a randomized control trial to caregivers of Veterans referred to home and community-based long-term care. Of primary interest is to examine whether participating in HI-FIVES leads to clinically significant increases in days spent at home for Veterans compared to caregivers in usual care. The investigators aim, through the training, to decrease the number of days over 12 months post-intervention that Veterans spend in the emergency department, hospital, or nursing home. Days spent in these settings reduces the Veteran's quality of life and increases health care costs to the VA. The investigators also will evaluate whether caregivers in HI-FIVES have clinically significant reductions in depressive symptoms post-intervention compared to caregivers in usual care.

DETAILED DESCRIPTION:
Anticipated Impacts on Veteran's Healthcare: Designing and implementing a training program for informal caregivers of functionally impaired Veterans (HI-FIVES) will enhance Veterans' ability to remain in their homes and satisfaction with care, as well as lower VA costs. Caregiver training can also improve caregiver wellbeing by alleviating feelings of depression and burden, which can also improve the care they provide to veterans. The investigators' caregiver training program is consistent with features of two recent national policy changes aimed to improve quality of care for veterans. First, providing training to informal caregivers of functionally impaired veterans is consistent with the 2000 Millennium Health Care Act, which mandated an unprecedented expansion in long-term care benefits to Veterans, and stipulated that, whenever possible, care be provided in the least restrictive environment possible-the home. Second, The Caregivers and Veterans Omnibus Health Services Act of 2010 mandated unprecedented support for informal caregivers of severely injured Operation Enduring Freedom/Operation Iraqi Freedom(OEF/OIF) Veterans, including providing caregiver training to informal caregivers of any era veteran. Achieving higher quality informal care supports both of these mandates. By partnering with VA providers, HI-FIVES will improve the skill of caregivers, thereby improving veteran health care quality and the ability for veterans to remain at home.

Project Background: Caregiver burnout, strain and burden are associated with caregiver depression and patient institutionalization. Furthermore, lack of skills among caregivers can lead to depression and anxiety as well as patient institutionalization. The investigators propose to evaluate an innovative program that supports and trains informal caregivers when veterans are referred to Veterans Health Administration (VHA) home and community-based care (HCBC), a critical moment in a veteran's VHA health care use trajectory. Referral to HCBC is a time when caregivers may face personal strain and uncertainty about demands involved in caregiving. As such, it presents a teachable moment to train caregivers to better meet the demands imposed by caregiving.

Project Objectives: To evaluate whether over 12 months, veterans with caregivers in the skill training program have clinically significant increases in days at home than veterans in usual care (e.g. days not in emergency department, hospital, or nursing home). In addition, the investigators will evaluate whether veterans in the skill training program have significantly lower VA costs of medical care or higher satisfaction with VHA over 6 and 12 months than veterans in usual care. Finally, the investigators will evaluate whether caregivers in the skill training program have clinically significant reductions in depressive symptoms, subjective burden, or increased satisfaction with VA healthcare at 6 and12 months than caregivers in usual care.

Project Methods: The study is a randomized controlled trial with data collection from caregiver-patient dyads before and after training, and at 6 and 12 months after program completion. Piloted in early 2012, the setting is the Social Work Service at the Durham VA Medical Center (VAMC). Patient inclusion criteria are patient referred to home and community-based services in the past 3 months, not eligible for hospice, residing at home, has an informal caregiver, and willing to let investigators contact the caregiver. Caregivers must be cognitively and physically capable to participate, understand English, not be treated for a substance abuse disorder, not be in another caregiver interventional study, and willing to participate in 3 phone call trainings and attend five group sessions at the VA. Caregivers in the control group will receive the training and support usually provided by HCBC and VA medical providers. To be referred successfully to HCBC, patients will have a minimum of 2 activity of daily living limitations, and are likely to have multimorbidity, including high rates of cognitive impairment (44% in the pilot). The target sample size will be 146 caregivers in each arm. Patient involvement will be limited to four short phone assessments (with mechanisms established for proxy respondents). Caregivers in the treatment arm will take part in three phone training sessions and five group sessions, and in both arms caregivers will be asked to provide four phone assessments. Descriptive statistics will be used to summarize all study variables. Of primary importance will be to examine the distribution of patient days spent at home during the first 3 months, the first 6 months, and over the entire 12 months of the post-intervention period (e.g. days not in ED, inpatient, or nursing home setting). Investigators will use the count-data regression model which best fits the investigators' data (Poisson, Negative Binomial or zero-inflated versions of Poisson or Negative Binomial) to test the primary hypothesis that veterans with caregivers in the skill training program will have significantly more days spent at home than veterans in usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to home and community-based services in the past 3 months,
* not eligible for hospice,
* residing at home,
* has an informal caregiver, and willing to let us contact the caregiver.

To be referred successfully to HCBC,

* patients will have a minimum of 2 activity of daily living limitations,
* and are likely to have multimorbidity, including high rates of cognitive impairment.

Exclusion Criteria:

* Cognitively impaired Caregiver
* Caregiver does not have access to a telephone.
* Severely impaired hearing or speech (Caregivers must be able to respond to phone calls).
* English Language Impaired - Caregiver
* Substance Abuse Disorders - Caregiver
* Caregiver participating in other caregiver intervention
* Patient referred only for physical or occupational therapy
* Patient or caregiver refuses informed consent
* Patient in hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van Houtven CH, Oddone EZ, Hastings SN, Hendrix C, Olsen M, Neelon B, Lindquist J, Weidenbacher H, Boles J, Chapman J, Weinberger M. Helping Invested Families Improve Veterans' Experiences Study (HI-FIVES): study design and methodology. Contemp Clin Trials. 2014 Jul;38(2):260-9. doi: 10.1016/j.cct.2014.05.003. Epub 2014 May 14. PMID 24837544
- [Derived] Shepherd-Banigan M, Smith VA, Lindquist JH, Cary MP Jr, Miller KEM, Chapman JG, Van Houtven CH. Identifying treatment effects of an informal caregiver education intervention to increase days in the community and decrease caregiver distress: a machine-learning secondary analysis of subgroup effects in the HI-FIVES randomized clinical trial. Trials. 2020 Feb 14;21(1):189. doi: 10.1186/s13063-020-4113-x. PMID 32059687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient's and their informal caregiver are randomized as a dyad to a single arm assignment, either HI-FIVES or Control.
Groups:
- Arm 1: Control - Caregivers: Caregivers in the control arm were referred to the VA Caregiver Support Program (usual care), as a resource for them as they care for the patient in the home.
  Helping Invested Families Improve Veterans Experiences Study - Control: Usual care was the Veteran patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. Caregivers in this arm were told about the caregiver support programs in the VHA and received the national VA caregiver hotline phone number. This mirrors efforts to support caregivers in the VA nationally.
- Arm 1: Control - Patients: The patient of each informal caregiver was also enrolled with contact limited to assessments.
  Helping Invested Families Improve Veterans Experiences Study - Control: Usual care was the Veteran patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. The patients in the usual care group were free to seek medical, psychological, social support, and social services available through VAMCs or any other source.
- Arm 2: HI FIVES - Caregivers: Caregivers took part in 3 phone training sessions and attended 4 group training sessions at the VA. They also had 2 post-group booster phone training sessions.
  Helping Invested Families Improve Veterans Experiences Study - HI FIVES: Caregivers received 3 individual calls with a nurse educator to address self-identified priority topics. These calls were tailored to the individual needs of Veteran-caregiver dyad. Caregivers then participated in evidence-based group sessions aimed to improve skills in clinical care, psychological care, and support-seeking. The curriculum was delivered by a trained nurse educator, the PI, and VA Caregiver Support staff. The 4 group training sessions were targeted to address common needs of Veterans and their caregivers. After the final group session, there were 2 follow-up booster calls at one and three months to check in with the caregiver.
- Arm 2: HI-FIVES - Patients: The patient of each informal caregiver was also enrolled with contact limited to assessments.
  Helping Invested Families Improve Veterans Experiences Study - HI-FIVES: Patients randomized to the HI-FIVES arm received no direct intervention. All intervention activities focused on the patient's informal caregiver. As with Usual care, patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. The patients in the HI-FIVES group were free to seek medical, psychological, social support, and social services available through VAMCs or any other source.
Period: Overall Study
Arm/Group | Arm 1: Control - Caregivers | Arm 1: Control - Patients | Arm 2: HI FIVES - Caregivers | Arm 2: HI-FIVES - Patients
Started | 123 | 123 | 119 | 119
Completed (Primary outcome is gathered from medical records. Survey outcomes have lower completion rates.) | 123 | 123 | 118 | 118
Not Completed | 0 | 0 | 1 | 1
Not completed — Dyad withdrew with data use prohibition | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: HI-FIVES - Caregivers: Caregivers took part in 3 phone training sessions and attended 4 group training sessions at the VA. They also had 2 post-group booster phone training sessions.
  Helping Invested Families Improve Veterans Experiences Study - HI FIVES: Caregivers received 3 individual calls with a nurse educator to address self-identified priority topics. These calls were tailored to the individual needs of Veteran-caregiver dyad. Caregivers then participated in evidence-based group sessions aimed to improve skills in clinical care, psychological care, and support-seeking. The curriculum was delivered by a trained nurse educator, the PI, and VA Caregiver Support staff. The 4 group training sessions were targeted to address common needs of Veterans and their caregivers. After the final group session, there were 2 follow-up booster calls at one and three months to check in with the caregiver.
- Arm 2: HI FIVES - Patients: The patient of each informal caregiver was also enrolled with contact limited to assessments.
  Helping Invested Families Improve Veterans Experiences Study - HI-FIVES: Patients randomized to the HI-FIVES arm received no direct intervention. All intervention activities focused on the patient's informal caregiver. As with Usual care, patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. The patients in the HI-FIVES group were free to seek medical, psychological, social support, and social services available through VAMCs or any other source.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control - Caregivers | Arm 1: Control - Patients | Arm 2: HI-FIVES - Caregivers | Arm 2: HI FIVES - Patients | Total
Number analyzed (Participants) | 123 | 123 | 119 | 119 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One enrolled patient/caregiver dyad in the intervention arm withdrew with an accompanying request to not use any of their data.
  years
    number analyzed (Participants) | 123 | 123 | 118 | 118 | 482
    (all) | 61.8 (12.60) | 72.9 (12.12) | 59.9 (11.78) | 73.7 (11.24) | 73.3 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One enrolled patient/caregiver dyad in the intervention arm withdrew with an accompanying request to not use any of their data.
  Participants
    number analyzed (Participants) | 123 | 123 | 118 | 118 | 482
    Female | 111 | 5 | 103 | 4 | 223
    Male | 12 | 118 | 15 | 114 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One enrolled patient/caregiver dyad in the intervention arm withdrew with an accompanying request to not use any of their data.
  Participants
    number analyzed (Participants) | 123 | 123 | 118 | 118 | 482
    Hispanic or Latino | 4 | 4 | 2 | 1 | 11
    Not Hispanic or Latino | 118 | 117 | 116 | 117 | 468
    Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One enrolled patient/caregiver dyad in the intervention arm withdrew with an accompanying request to not use any of their data.
  Participants
    number analyzed (Participants) | 123 | 123 | 118 | 118 | 482
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
    Asian | 1 | 1 | 0 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Black or African American | 59 | 60 | 50 | 48 | 217
    White | 48 | 48 | 56 | 60 | 212
    More than one race | 15 | 13 | 11 | 9 | 48
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: One enrolled patient/caregiver dyad in the intervention arm withdrew with an accompanying request to not use any of their data.
  Participants
    United States: number analyzed (Participants) | 123 | 123 | 118 | 118 | 482
    United States | 123 | 123 | 118 | 118 | 482

OUTCOME MEASURES:

1. Primary Outcome: Patient Days in the Community (e.g. Days Not in Emergency Department, Inpatient, or Nursing Home Setting)
Description: Days at home is defined as the total numbers of days of VA, inpatient and post-acute facility care subtracted from 365 (or number of days living in 12 month post randomization period if deceased). Mean was estimated using a generalized linear model.
Time Frame: 12 months
Population: All enrolled subjects were included in the analysis of the primary outcome, except for the one subject who withdrew permission to use data.
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- Arm 1: Control: Caregivers in the control arm were referred to the VA Caregiver Support Program (usual care), as a resource for them as they care for the patient in the home. The patient of each caregiver was also enrolled with contact limited to assessments.
  Helping Invested Families Improve Veterans Experiences Study - Control: Usual care was the Veteran patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. The patients in the usual care group were free to seek medical, psychological, social support, and social services available through VAMCs or any other source. In addition, caregivers in this arm were told about the caregiver support programs in the VHA and received the national VA caregiver hotline phone number. This mirrors efforts to support caregivers in the VA nationally.
- Arm 2: HI FIVES: Caregivers took part in 3 phone training sessions and attended 4 group training sessions at the VA. They also had 2 post-group booster phone training sessions. The patient of each caregiver was also enrolled with contact limited to assessments.
  Helping Invested Families Improve Veterans Experiences Study - HI FIVES: Caregivers received 3 individual calls with a nurse educator to address self-identified priority topics. These calls were tailored to the individual needs of Veteran-caregiver dyad. Caregivers then participated in evidence-based group sessions aimed to improve skills in clinical care, psychological care, and support-seeking. The curriculum was delivered by a trained nurse educator, the PI, and VA Caregiver Support staff. The 4 group training sessions were targeted to address common needs of Veterans and their caregivers. After the final group session, there were 2 follow-up booster calls at one and three months to check in with the caregiver.
Arm/Group | Arm 1: Control | Arm 2: HI FIVES
Number analyzed (Participants) | 123 | 118
days | 352.87 [348.76 to 355.94] | 353.62 [349.75 to 356.51]

2. Secondary Outcome: Total Costs to the VA
Description: VA utilization costs will be summarized across VA and non-VA contracted care and will capture all outpatient costs (laboratory, radiology, pharmacy, surgery, nursing, and treat and release ED visits) and inpatient costs (similar categories). Mean was estimated using a generalized linear model.
Time Frame: 12 months
Population: All enrolled patient subjects were included in the analysis of this outcome, except for the one subject who withdrew permission to use data.
Measure: Mean (95% Confidence Interval); unit: Dollars
Arm/Group | Arm 1: Control | Arm 2: HI FIVES
Number analyzed (Participants) | 123 | 118
Dollars | 44227.55 [34772.66 to 56253.30] | 41157.17 [33455.72 to 50631.47]

3. Secondary Outcome: Satisfaction With Healthcare
Description: Consumer Assessment of Healthcare Providers and Systems (CAHPS). Used by the VA Office of Performance and Quality, this outcome is considered a key measure of patient satisfaction with inpatient and outpatient care. The investigators will focus on a global satisfaction measure about the health plan: "Using any number from 0 to 10, where 0 is the worst health care possible and 10 is the best health care possible, what number would [PATIENT: you/the patient (if not competent to answer for themselves) use to rate all of your/his/her] [CAREGIVER: you use to rate all the patient's] health care in the VA in the last 3 months?" This measure was asked of both the patient and their informal caregiver. If the patient was not competent to answer for themselves, the caregiver was asked to respond on the patient's behalf. Mean was estimated using a linear mixed model.
Time Frame: 3 months
Population: This measure was collected from both the patient (or their proxy if not competent) and their informal caregiver. We had one dyad who withdrew from Arm 2 (HI FIVES) and asked us not to use their data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Arm 1: Control (CAREGIVER): Caregivers in the control arm were referred to the VA Caregiver Support Program (usual care), as a resource for them as they care for the patient in the home.
  Helping Invested Families Improve Veterans Experiences Study - Control: Usual care was the Veteran patient care and caregiver support normally offered once the Geriatrics and Extended Care (GEC) referral process has occurred. This entails the patient and caregiver work with the assigned social worker to obtain home and community based care (HCBC) services. The patients in the usual care group were free to seek medical, psychological, social support, and social services available through VAMCs or any other source. In addition, caregivers in this arm were told about the caregiver support programs in the VHA and received the national VA caregiver hotline phone number. This mirrors efforts to support caregivers in the VA nationally.
- Arm 1: Control (PATIENT); Arm 2: HI FIVES (PATIENT): The patient of each caregiver was also enrolled with contact limited to assessments.
- Arm 2: HI FIVES (CAREGIVER): Caregivers took part in 3 phone training sessions and attended 4 group training sessions at the VA. They also had 2 post-group booster phone training sessions.
  Helping Invested Families Improve Veterans Experiences Study - HI FIVES: Caregivers received 3 individual calls with a nurse educator to address self-identified priority topics. These calls were tailored to the individual needs of Veteran-caregiver dyad. Caregivers then participated in evidence-based group sessions aimed to improve skills in clinical care, psychological care, and support-seeking. The curriculum was delivered by a trained nurse educator, the PI, and VA Caregiver Support staff. The 4 group training sessions were targeted to address common needs of Veterans and their caregivers. After the final group session, there were 2 follow-up booster calls at one and three months to check in with the caregiver.
Arm/Group | Arm 1: Control (CAREGIVER) | Arm 1: Control (PATIENT) | Arm 2: HI FIVES (CAREGIVER) | Arm 2: HI FIVES (PATIENT)
Number analyzed (Participants) | 123 | 123 | 118 | 118
units on a scale | 8.29 [7.97 to 8.61] | 8.09 [7.70 to 8.48] | 8.58 [8.25 to 8.89] | 8.38 [7.99 to 8.77]

4. Secondary Outcome: Caregiver Depressive Symptoms
Description: The investigators selected the Center for Epidemiological Studies-Depression 10 scale (CESD-10) measure of depressive symptoms because the respondent burden is low and in order to maximize comparability with REACH I and REACH II. Range is 0-30 with a higher score indicates greater depressive symptoms. Mean was estimated using a linear mixed model.
Time Frame: 3 months
Population: All enrolled caregiver subjects were included in the analysis of this outcome, except for the one dayd who withdrew permission to use data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Control | Arm 2: HI FIVES
Number analyzed (Participants) | 123 | 118
units on a scale | 8.95 [7.90 to 10.00] | 8.75 [7.69 to 9.82]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of enrollment up to 365 days post-randomization.
Description: We systematically collected adverse event reports for the patient participants as we collected all medical records, both VA and non-VA, for the duration of their enrollment. We collected adverse event reports from the caregivers on a self-reported, non-systematic, basis.
Arm/Group | Arm 1: Control - Caregivers | Arm 1: Control - Patients | Arm 2: HI-FIVES - Caregivers | Arm 2: HI FIVES - Patients
All-Cause Mortality (participants affected / at risk) | 0/123 | 10/123 | 0/118 | 14/118
Serious Adverse Events (participants affected / at risk) | 0/123 | 71/123 | 0/118 | 68/118
Other Adverse Events (participants affected / at risk) | 0/123 | 60/123 | 0/118 | 57/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control - Caregivers (N=123) | Arm 1: Control - Patients (N=123) | Arm 2: HI-FIVES - Caregivers (N=118) | Arm 2: HI FIVES - Patients (N=118)
Death (Cardiac disorders) | NA | 0 (0) | NA | 2 (2)
Death (General disorders) | NA | 5 (5) | NA | 3 (3)
Death (Injury, poisoning and procedural complications) | NA | 0 (0) | NA | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 2 (2) | NA | 1 (1)
Death (Nervous system disorders) | NA | 2 (2) | NA | 3 (3)
Death (Renal and urinary disorders) | NA | 0 (0) | NA | 1 (1)
Death (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | NA | 3 (3)
Hospitalization (Blood and lymphatic system disorders) | NA | 1 (1) | NA | 3 (3)
Hospitalization (Cardiac disorders) | NA | 11 (15) | NA | 9 (10)
Hospitalization (Endocrine disorders) | NA | 3 (4) | NA | 2 (2)
Hospitalization (Gastrointestinal disorders) | NA | 6 (11) | NA | 3 (4)
Hospitalization (General disorders) | NA | 10 (11) | NA | 4 (5)
Hospitalization (Infections and infestations) | NA | 15 (20) | NA | 14 (19)
Hospitalization (Injury, poisoning and procedural complications) | NA | 12 (13) | NA | 6 (7)
Hospitalization (Metabolism and nutrition disorders) | NA | 1 (1) | NA | 3 (3)
Hospitalization (Musculoskeletal and connective tissue disorders) | NA | 4 (4) | NA | 2 (2)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 2 (2) | NA | 2 (2)
Hospitalization (Nervous system disorders) | NA | 10 (11) | NA | 8 (8)
Hospitalization (Renal and urinary disorders) | NA | 4 (5) | NA | 10 (12)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | NA | 12 (19) | NA | 12 (14)
Hospitalization (Skin and subcutaneous tissue disorders) | NA | 1 (1) | NA | 1 (1)
Hospitalization (Surgical and medical procedures) | NA | 4 (5) | NA | 14 (16)
Hospitalization (Vascular disorders) | NA | 4 (6) | NA | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control - Caregivers (N=123) | Arm 1: Control - Patients (N=123) | Arm 2: HI-FIVES - Caregivers (N=118) | Arm 2: HI FIVES - Patients (N=118)
ED Visit (Gastrointestinal disorders) | NA | 13 (17) | NA | 8 (13)
ED Visit (General disorders) | NA | 6 (7) | NA | 12 (12)
ED Visit (Infections and infestations) | NA | 19 (24) | NA | 9 (12)
ED Visit (Injury, poisoning and procedural complications) | NA | 17 (18) | NA | 22 (34)
ED Visit (Musculoskeletal and connective tissue disorders) | NA | 21 (29) | NA | 17 (20)
ED Visit (Nervous system disorders) | NA | 5 (5) | NA | 6 (7)
ED Visit (Respiratory, thoracic and mediastinal disorders) | NA | 6 (7) | NA | 2 (2)
ED Visit (Vascular disorders) | NA | 12 (17) | NA | 12 (13)

LIMITATIONS AND CAVEATS:
HI-FIVES was tested in a single VA medical center. It was likely underpowered to detect statistically significant differences in primary outcome due to greater than expected variance. A larger sample size may be needed to detect true differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes